CLINICAL TRIAL: NCT06763666
Title: A Multicenter, Prospective, Randomized Controlled Study Comparing the Efficacy and Safety of CLAG(Cladribine, Cytarabine and G-CSF) Combined With Venetoclax and CLAG in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: CLAG+VEN vs CLAG in the Treatment of Relapsed/Refractory AML
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou No.12 People's Hospital (Other Government); Guangzhou Panyu Central Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangzhou First People's Hospital (Other); Foresea Life Insurance Guangzhou General Hospital (Unknown); Guangdong Second Provincial General Hospital (Other); Jiangmen Central Hospital (Other); Shantou Central Hospital (Other); Maoming People's Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Hainan General Hospital (Other); Dongguan People's Hospital (Other Government); Tungwah Hospital of Sun Yat-Sen University (Unknown); Shenzhen Hospital of Southern Medical University (Other); Central People's Hospital of Zhanjiang (Other); ZhuHai Hospital (Other); Shenzhen Second People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); LiuZhou People's Hospital (Other); First People's Hospital of Foshan (Other); Southern Medical University, China (Other); Affiliated Hospital of Guangdong Medical University (Other); Guilin Medical University, China (Other); Yuebei People's Hospital (Other); Huizhou Municipal Central Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-639
Record Dates: First submitted 2024-12-30; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Granulocyte Colony-Stimulating Factor; Filgrastim; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLAGV regimen (Experimental): CLAG combined with venetoclax for relapsed/refractory AML. Patients were randomized and those entering the experimental group received cladribine, cytarabine, G-CSF and venetoclax.
  Venetoclax is administered orally at 400mg/d on days 2-8. When combination with P450 3A4 inhibitor, VEN should be reduced to 100-200mg/d and monitoring of VEN blood concentrations is recommended at qualified centers. Cladribine is administered intravenously at a dose of 5 mg/m2/d on days 1-5. Cytarabine is administered intravenously at a dose of 1g/m2/d on days 1-5, starting 2h after cladribine and maintained for more than 3h. The dose of G-CSF was 5ug/kg/d subcutaneously injected on days 0-5. Generally, starting 12 hours before the start of chemotherapy, if the absolute value of white blood cell count is ≥ 20×10^9/L, the use is suspended.For patients with FLT3 mutations, corresponding inhibitors such as sorafenib and gilteritinib can be combined.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: G-CSF; Drug: Venetoclax
- CLAG regimen (Active Comparator): CLAG regimen for relapsed/refractory AML. Patients were randomized and those entering the experimental group received cladribine, cytarabine, G-CSF.
  Cladribine is administered intravenously at a dose of 5 mg/m2/d on days 1-5. Cytarabine is administered intravenously at a dose of 1g/m2/d on days 1-5, starting 2h after cladribine and maintained for more than 3h. The dose of G-CSF was 5ug/kg/d subcutaneously injected on days 0-5. Generally, starting 12 hours before the start of chemotherapy, if the absolute value of white blood cell count is ≥ 20×10^9/L, the use is suspended.For patients with FLT3 mutations, corresponding inhibitors such as sorafenib and gilteritinib can be combined.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: G-CSF

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; CdA
Drug: Cytarabine — Given IV
  Other Names: Ara-C
Drug: G-CSF — Given SC
  Other Names: Filgrastim; Granulocyte Colony-stimulating Factor
Drug: Venetoclax — Given PO
  Other Names: Venclexta
  Arms: CLAGV regimen

SUMMARY:
This is a multicenter, prospective, randomized controlled clinical study comparing the efficacy and safety of CLAG+VEN and CLAG regimens in relapsed/refractory(r/r) AML.

DETAILED DESCRIPTION:
The efficacy and prognosis of relapsed/refractory(r/r) AML are very poor, and there is no standard chemotherapy regimen were defined for r/r AML. Cladribine, a purine analogue, exerts cytotoxic, proapoptotic, and antiproliferative effects on AML cells. Previous studies have confirmed the efficacy of cladribine in the treatment of r/r AML, with a response rate of 30-45%.Our previous experience has shown that CLAG in combination of venetoclax are effective with tolerable toxicity profiling. However, there is a lack of multicenter, prospective, randomized controlled trials to further confirm the results. Therefore, a clinical study is planned to evaluate the efficacy and safety of CLAG+VEN compared to CLAG in r/r AML who were eligible for intensive therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of AML according to the World Health Organization (WHO) classification.
2. All patients should aged 18 to 65 years.
3. Diagnosed of relapsed and refractory AML, according to The guidelines for diagnosis and treatment of relapse /refractory acute myelogenous leukemia in China（2023）
4. Diagnostic criteria for relapsed AML: Leukemia cells reappear in the peripheral blood or primitive cells in the bone marrow ≥ 5% (excluding other reasons such as bone marrow regeneration after consolidation chemotherapy) after CR, or leukemia cell infiltration appears outside the marrow.
5. Diagnostic criteria for refractory AML: The newly diagnosed patients who failed to respond to two courses of standard treatment; Patients who relapsed within 12 months after consolidation intensive therapy; Patients who relapsed after 12 months and failed to respond to conventional chemotherapy; Patients with two or more recurrences; Patients with persistent extramedullary leukemia.
6. The score of Eastern Cooperative Oncology Group (ECOG) is 0-2.
7. Renal function: creatinine clearance rate ≥ 30ml/min.
8. Liver function: ALT<5 times normal value, bilirubin<3 times normal value.
9. Predicted survival ≥ 3 months.
10. Able to accept oral Venetoclax.
11. Sign an informed consent form and be able to understand and follow the procedures required by this protocol.

Exclusion Criteria:

1. Diagnosed of acute promyelocytic leukemia (AML-M3)
2. Patients with central nervous system (CNS) invasion.
3. Cardiac function < grade 2.
4. Known human immunodeficiency virus (HIV) infection.
5. Other clinically significant uncontrolled conditions, including but not limited to: a. uncontrolled or active systemic infections (viruses, bacteria, or fungi); b. Chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) requiring treatment; c. Secondary tumors requiring active treatment.
6. Allergy to experimental drugs.
7. Pregnant and lactating women.
8. Patients who ineligible for the study according to the investigator's assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite Complete remission (cCR, CR+CRi) | At the end of Cycle 1 (each cycle is 28 days)
  Will compare composite complete remission(CR+CRi: complete response [CR] and complete response with incomplete blood count recovery [CRi]) between CLAGV regimen and CLAG regimen

SECONDARY OUTCOMES:
Overall Response rate (ORR) | At the end of Cycle 1 (each cycle is 28 days)
  Will compare ORR(completed remission[CR], completed remission with incomplete blood count recovery[CRi], and partial remission[PR]) rates between the study arms
MRDneg CR rate | At the end of Cycle 1 (each cycle is 28 days)
  Will compare MRD-negative cCR rates between the study arms
Overall Survival(OS) | 1 year post treatment
  Will compare OS between the study arms
Relapse free survival(RFS) | 1 year post treatment
  Will compare RFS between the study arms
Duration of completed response(DoR) | 1 year post treatment
  Will compare DoR between the study arms
Relapse rate | 1 year post treatment
  Will compare relapse rate between the study arms
Incidence of Adverse Events | Duration of treatment, up to 1 year
  Will use the CTCAE (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events) version 5.0 for toxicity and adverse event reporting. Will describe the incidence of infection and treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Guopan Yu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No